CLINICAL TRIAL: NCT00367991
Title: Effects of Recombinant Human Erythropoietin on Platelet Function in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0506000140; 0555844T
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2017-12

CONDITIONS: Myocardial Infarction
Keywords: Platelet function tests; Erythropoietin; Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): recombinant human erythropoietin 200 U/kg IV daily for 3 days
  Interventions: Drug: Recombinant human erythropoietin alfa (drug)
- B (Placebo Comparator): Normal saline volume to match active treatment IV daily for 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant human erythropoietin alfa (drug) — 200 U/kg IV daily for 3 days vs. matched volume of normal saline IV daily for 3 days
  Arms: A
Drug: Placebo — Normal saline to match active drug (rHuEpo)
  Arms: B

SUMMARY:
The purpose of this study is to see if a naturally-occurring hormone called erythropoietin changes the action of platelets in the blood. Patients with heart attacks are treated with medicines to reduce the clotting action of platelets. This study is trying to determine whether erythropoietin alters the clotting action of platelets in patients receiving anti-platelet medicines. It is important to understand the effects of erythropoietin on platelets since preliminary studies in animals suggest that erythropoietin may protect the heart from damage during a heart attack.

DETAILED DESCRIPTION:
Anti-apoptotic effects of erythropoietin in experimental myocardial infarction (MI) and ischemia-reperfusion injury suggest potential for therapeutic benefit in patients with acute MI. Before the therapeutic potential of recombinant human erythropoietin (rHuEpo) in acute MI can be tested in large clinical trials, more information on the effects of short-term rHuEpo on platelet function are needed. Accordingly, the current proposal aims to determine the effects of rHuEpo (at a dose previously shown not to inhibit the anti-platelet effects of aspirin and clopidogrel in healthy subjects) on platelet function and other safety measures and measure of infarct size in patients with acute coronary syndromes receiving clinically-indicated standard anti-platelet therapy with aspirin, clopidogrel and glycoprotein Iib-IIIa inhibitors.

Specific Aim 1: To determine the effects of intravenous rHuEpo 400 U/kg daily for 3 days vs. placebo on in vivo and in vitro platelet function in patients with acute MI undergoing percutaneous revascularization.

Specific Aim 2: To obtain pilot data to estimate the effects of administration of rHuEpo 400 U/kg daily for 3 days vs. placebo on biochemical markers of myocardial infarction size and left ventricular ejection fraction in patients with acute MI undergoing percutaneous revascularization

ELIGIBILITY:
Inclusion Criteria:

* Age 21-75 years
* Clinical evidence of acute myocardial infarction (MI) with total or sub-total occlusion on angiogram
* Status post percutaneous revascularization procedure for acute MI with TIMI 3 flow
* Ongoing clinically-indicated treatment with aspirin, thienopyridines

Exclusion Criteria:

* Hemodynamic instability/shock or severe congestive heart failure
* Time from onset of chest pain to revascularization procedure > 16 hours
* Use of intravenous thrombolytic agents for treatment of MI
* Known need for additional revascularization procedures

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Katz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Result] Tang YD, Hasan F, Giordano FJ, Pfau S, Rinder HM, Katz SD. Effects of recombinant human erythropoietin on platelet activation in acute myocardial infarction: results of a double-blind, placebo-controlled, randomized trial. Am Heart J. 2009 Dec;158(6):941-7. doi: 10.1016/j.ahj.2009.06.032. PMID 19958860

RESULTS

PARTICIPANT FLOW:
Groups:
- rHuEPO: recombinant human erythropoietin 200 U/kg IV daily for 3 days
- Placebo: Normal saline volume to match active treatment IV daily for 3 days
Period: Overall Study
Arm/Group | rHuEPO | Placebo
Started | 29 | 15
Completed | 27 | 13
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rHuEPO | Placebo | Total
Number analyzed (Participants) | 29 | 15 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 13 | 35
  >=65 years | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12) | 53 (9) | 56 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 21 | 10 | 31
Region of Enrollment [Number; unit: participants]
  United States | 29 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Time
Description: An integrated measure of in vivo platelet function and tissue hemostasis.
Time Frame: Change from Day 3 to Day 10
Population: ITT
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- Placebo: normal saline
- rHuEPO: recombinant human erythropoietin
Arm/Group | Placebo | rHuEPO
Number analyzed (Participants) | 15 | 29
seconds | 1020 [960 to 1110] | 1020 [960 to 1110]

2. Primary Outcome: Platelet Function Assay Closure Time
Time Frame: Change from Day 3 to Day 10
Population: ITT
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Placebo | rHuEPO
Number analyzed (Participants) | 15 | 29
seconds | 251 [185 to 301] | 281 [173 to 301]

3. Secondary Outcome: Left Ventricular Ejection Fraction
Time Frame: Day 1 and Day 10
Population: These data were not collected due to lack of funds.
Arm/Group | Placebo | rHuEPO
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Serum Markers of Myocyte Damage
Description: Myocyte Damage is represented by Creatine phosphokinase (CPK). CPK is measured in U/L, as scalar measure of the enzyme activity. CPK was measured for clinical indications laboratory.
Time Frame: Baseline
Population: ITT
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Placebo | rHuEPO
Number analyzed (Participants) | 15 | 29
U/L | 817 [114 to 2040] | 652 [379 to 868]

5. Secondary Outcome: Circulating Endothelial Progenitor Cells
Time Frame: Day 3 and Day 10
Population: Endothelial progenitor cells could not be isolated and are therefore not reported.
Arm/Group | Placebo | rHuEPO
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Serum Markers of Apoptosis
Description: Apoptosis is represented by Fas ligand (FasL or CD95L). FasL (CD95L) is measured in pg/mL.
Time Frame: Day 1 and Day 10
Population: ITT
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | rHuEPO
Number analyzed (Participants) | 15 | 29
pg/mL
  Day 1 | 45 (12) | 56 (19)
  Day 10 | 60 (18) | 63 (22)

ADVERSE EVENTS:
Arm/Group | rHuEPO | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/15
Other Adverse Events (participants affected / at risk) | 0/29 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rHuEPO (N=29) | Placebo (N=15)
hospitalization (Cardiac disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No